CLINICAL TRIAL: NCT06757075
Title: A Comparison of Standard Dose of Ibuprofen Alone, Alternating, or Combined With Acetaminophen for the Management of Postoperative Discomfort in Young Children Following Dental Rehabilitation Under General Anesthesia
Brief Title: Management of Postoperative Discomfort in Young Children Following Dental Rehabilitation Under General Anesthesia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Franciscan Hospital For Children, INC. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-001FC
Record Dates: First submitted 2024-12-24; First posted 2025-01-03 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Pain, Postoperative
Keywords: Dental rehabilitation under general anesthesia (DRGA); Dental surgery patients 4-6 years; Acetominophen; Ibuprofen; Pacing analgesics
MeSH Terms: conditions — Pain, Postoperative | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Alternating analgesics (Experimental): Participants randomized into this arm will be given alternating Ibuprofen and Acetaminophen every 6 hours, alternating the two medications every 3 hours: first dose ibuprofen, three hours later acetaminophen for 24 hours.
  Interventions: Drug: Ibuprofen; Drug: Acetominophen
- Simultaneous post-operative analgesics (Experimental): Participants randomized into this arm will be given simultaneous Ibuprofen and Acetaminophen every 6 hours for 24 hours.
  Interventions: Drug: Ibuprofen; Drug: Acetominophen
- Control Standard of Care (Active Comparator): Participants randomized into this arm will be given Ibuprofen every 6 hours for 24 hours.
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — 10 mg/kg/dose of ibuprofen will be given every 6 hours for 24 hours post surgery
  Other Names: Motrin
Drug: Acetominophen — 15 mg/kg/dose of acetominophen will be given every 6 hours for 24 hours post surgery
  Other Names: Tylenol
  Arms: Alternating analgesics; Simultaneous post-operative analgesics

SUMMARY:
The purpose of this study is to investigate the effectiveness of various oral analgesic regimens in minimizing post-operative pain and discomfort in young children following dental rehabilitation under general anesthesia (DRGA). In this randomized controlled trial, three analgesic regimens following DRGA in Franciscan Children's Hospital will be compared using both self-report and behavioral measures.

The analgesic therapies to be investigated are ibuprofen monotherapy, alternating ibuprofen and acetaminophen dual-therapy, and combined ibuprofen and acetaminophen dual-therapy. For the purposes of this study, combined therapy is defined as the simultaneous administration of acetaminophen and ibuprofen at regular intervals, whereas alternating therapy is defined as one analgesic (acetaminophen or ibuprofen) administered within a 3 hour interval of the other.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I-II
* Requiring Oral Rehabilitation under General Anesthesia
* Possess legal guardians proficient in English
* Not have a history of any adverse/allergic reaction to nonsteroidal anti-inflammatory drugs (NSAIDs) or Acetaminophen

Exclusion Criteria:

* ASA III or IV
* Asthma diagnosis
* Contraindication to acetaminophen or ibuprofen

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Dental discomfort assessed by the abbreviated DDQ-8 | day of surgery, one pay post surgery, 2 days post surgery, 15 days post surgery
  The Dental Discomfort Questionnaire (DDQ-8)-Abbreviated is an 8 item questionnaire completed by the caregiver. Responses to each question are Yes=2 and No=0 creating a possible range of total scores of 0-16 with higher scores correlated with more dental discomfort.
Pain assessment based on the FLACC | day of surgery, one pay post surgery, 2 days post surgery, 15 days post surgery
  The Face, Legs, Activity, Cry, and Consolability (FLACC) scale assesses pain by the caregiver on 5 aspects of behavior: (F) facial expression; (L) leg movement; (A) activity; (C) cry; (C) consolability. Each behavior is rated 0 to 2 resulting in a range of scores from 0 to 10 with higher scores correlated with more pain.

CONTACTS AND LOCATIONS:
Overall Officials: Keri Discepolo, DDS MPH, Principal Investigator — BU Goldman School of Dental Medicine, Pediatrics
Locations (1):
- Franciscan Children's Hospital, Brighton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No